CLINICAL TRIAL: NCT07381374
Title: Study Protocol for a Randomized Controlled of Fecal Microbiota Transplantation Via Different Routes in Children With Moderate-to-Severe Autism Spectrum Disorder
Brief Title: Fecal Microbiota Transplantation in Children With ASD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Children's Hospital (Other Government)
Collaborators: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other); Shenzhen Medical Academy of Research and Translation (Unknown)
Responsible Party: Principal Investigator, Dongling Dai, Professor, Shenzhen Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202500102
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Fecal Microbiota Transplantation; Microbiome; children
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (FMT-NJT) (Active Comparator): active FMT via nasojejunal tube + sham colonoscopy
  Interventions: Procedure: ctive FMT via Nasojejunal Tube (FMT-Upper GI)
- Group 2 (FMT-C) (Active Comparator): active FMT via colonoscopy with placement of a transendoscopic enteral tube (TET) secured at the cecum during the first session, followed by two subsequent infusions via the indwelling TET + sham nasojejunal intubation.
  Interventions: Procedure: Active FMT via Colonoscopy and Transendoscopic Tube (FMT-Lower GI)
- Group 3 (Control) (Placebo Comparator): placebo via nasojejunal tube + placebo via colonoscopy (sham procedures for both routes)
  Interventions: Procedure: Placebo via Sham Procedures (Sham-Control)

INTERVENTIONS:
Procedure: ctive FMT via Nasojejunal Tube (FMT-Upper GI) — Intervention: Active FMT via Nasojejunal Tube (FMT-Upper GI) Intervention Type: Procedure + Biological Intervention Name: Upper Gastrointestinal-Targeted Fecal Microbiota Transplantation Description: Participants in this group receive active fecal microbiota suspension delivered to the jejunum (upper gastrointestinal tract). Under endoscopic guidance, a nasojejunal tube is placed with its tip positioned past the Ligament of Treitz. The active FMT preparation is then infused slowly through this tube. Additionally, participants undergo a sham colonoscopy (simulated procedure under anesthesia where the scope is inserted to the rectosigmoid junction with minimal water/air insufflation, but no FMT is administered).
  Dosage: 5 mL per kilogram of body weight, with a maximum total volume of 100 mL per infusion.
  Frequency: Administered once every other day, for a total of three sessions over 5 days.
  Arms: Group 1 (FMT-NJT)
Procedure: Active FMT via Colonoscopy and Transendoscopic Tube (FMT-Lower GI) — Participants in this group receive active fecal microbiota suspension delivered to the cecum (lower gastrointestinal tract). The intervention involves two phases:
  First Session (Day 0): Under general anesthesia, a full colonoscopy is performed to reach the cecum. The active FMT preparation is infused directly into the cecum. Subsequently, a transendoscopic enteral tube (TET) is advanced through the colonoscope and its tip is secured in the cecum using endoscopic clips.
  Second & Third Sessions (Days 2 & 4): The active FMT preparation is infused through the indwelling TET at the bedside, without the need for repeat colonoscopy or general anesthesia.
  Additionally, participants undergo a sham nasojejunal intubation (a tube is placed into the stomach and secured, and a placebo is infused).
  Dosage: 5 mL per kilogram of body weight, with a maximum total volume of 100 mL per infusion.
  Frequency: Administered once every other day, for a total of three sessions over 5 days.
  Arms: Group 2 (FMT-C)
Procedure: Placebo via Sham Procedures (Sham-Control) — Participants in this control group undergo both sham procedures with infusion of an inactivated placebo suspension, which is visually and physically identical to the active FMT preparation but contains no viable microbiota.
  Sham Nasojejunal Intubation: A tube is placed into the stomach (not the jejunum) and secured. The placebo suspension is infused.
  Sham Colonoscopy: Under anesthesia, a simulated colonoscopy is performed (scope inserted to rectosigmoid junction with minimal insufflation). No substance is infused during this sham procedure.
  This double-sham design ensures that both potential delivery routes are "simulated" for the control group.
  Dosage: Volume-matched to the active FMT arms (5 mL/kg, max 100 mL) for the nasogastric infusion. No infusion during sham colonoscopy.
  Frequency: The placebo infusion (during sham NJ intubation) occurs once every other day, for a total of three sessions over 5 days, coinciding with the two sham procedures.
  Arms: Group 3 (Control)

SUMMARY:
This is a single-center, randomized, double-dummy, triple-blind, placebo-controlled, three-arm parallel-group superiority trial. The study aims to compare the efficacy and safety of Fecal Microbiota Transplantation (FMT) administered via two different invasive routes-nasojejunal tube (NJT) and colonoscopy-versus a placebo control in children aged 3-16 years with moderate-to-severe Autism Spectrum Disorder (ASD). A total of 75 participants will be randomized in a 1:1:1 ratio to receive either active FMT via NJT with sham colonoscopy, active FMT via colonoscopy with sham NJT, or placebo via both routes. All participants will continue their stable behavioral interventions throughout the study. The primary outcome is the change from baseline to Week 24 in the total score of the Childhood Autism Rating Scale (CARS). Secondary outcomes include changes in other behavioral and gastrointestinal symptom scores, gut microbiota profiling, and safety assessments over 48 weeks.

DETAILED DESCRIPTION:
Background:

Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder often accompanied by gastrointestinal (GI) symptoms and gut microbiota dysbiosis. Fecal Microbiota Transplantation (FMT) has shown promise in modulating the gut-brain axis and improving both behavioral and GI symptoms in preliminary ASD studies. However, the optimal route of FMT administration remains unclear, and high-quality comparative evidence is lacking.

Objectives:

Primary: To compare the efficacy of FMT delivered via NJT versus colonoscopy versus placebo in improving social interaction and communication, as measured by the change in CARS total score from baseline to Week 24.

Secondary: To evaluate effects on social responsiveness (SRS), aberrant behaviors (ABC), sensory processing (SSP), sleep quality (CSHQ), GI symptoms (GSRS), gut microbiota engraftment dynamics, and safety/tolerability.

Methods:

Design: Single-center, randomized, double-dummy, triple-blind, placebo-controlled, three-arm parallel-group trial.

Participants: 75 children aged 3-16 years with DSM-5-confirmed moderate-to-severe ASD (CARS ≥36) and stable behavioral intervention.

Interventions:

Group 1 (FMT-NJT): Active FMT via NJT + sham colonoscopy. Group 2 (FMT-C): Active FMT via colonoscopy with placement of a transendoscopic enteral tube (TET) in the cecum for subsequent infusions + sham NJT.

Group 3 (Control): Placebo via both NJT and colonoscopy (sham procedures). Dosage: 5 mL/kg (max 100 mL) per infusion, administered every other day for three sessions.

Blinding: Triple-blind-participants/guardians, outcome assessors, and data analysts are blinded. An independent pharmacy unit prepares identical active and placebo preparations.

Assessments: Behavioral scales (CARS, SRS, ABC, SSP, CSHQ), GI symptoms (GSRS), stool metagenomics, and safety monitoring at baseline, Weeks 2, 6, 12, 24, and 48.

Sample Size: 25 per group (total N=75), calculated to detect a 2.5-point difference in CARS change with 80% power, accounting for 15% dropout.

Randomization: Centralized block randomization stratified by age and baseline CARS severity.

Statistical Analysis: ANCOVA for primary outcome with baseline adjustment; mixed models for repeated measures; descriptive and inferential methods for secondary and safety outcomes.

Outcomes:

Primary: Change in CARS total score from baseline to Week 24. Secondary: Changes in SRS, ABC, GSRS, SSP, CSHQ scores; microbiota composition/function; incidence and severity of adverse events (CTCAE v5.0).

Significance: This trial will provide high-level evidence on whether the therapeutic effect of FMT in ASD depends on the gastrointestinal delivery site. The novel TET-based protocol for repeated cecal delivery allows for a rigorous comparison of microbial engraftment in the lower versus upper GI tract. The results will guide the optimization of microbiota-targeted therapies for ASD and other conditions linked to the gut-brain axis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3-16 years.
* Diagnosed with ASD according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), with a Childhood Autism Rating Scale (CARS) total score ≥36 (moderate-to-severe autism).
* Legal guardians fully comprehend the trial's informed consent and voluntarily provide written consent.
* Compliance with follow-up visits, examinations, and specimen collection.
* No probiotic supplements consumed within the preceding 3 months.

Exclusion Criteria:

* Use of probiotics or prebiotics within 3 months prior to enrollment.
* Antibiotic usage within 1 month prior to enrollment.
* Presence of fever (axillary temperature ≥37.5°C).
* Dependency on tube feeding.
* Severe gastrointestinal conditions requiring immediate intervention (e.g., life-threatening intestinal obstruction, perforation, hemorrhage, ulcerative colitis, Crohn's disease, celiac disease, or eosinophilic esophagitis).
* Diagnosis of severe malnutrition, underweight status (BMI-for-age <3rd percentile), or severe immunodeficiency disorders.
* History of severe allergic reactions (e.g., anaphylaxis).
* Monogenic disorders (e.g., Fragile X syndrome, Rett syndrome).
* Comorbid psychiatric diagnoses, including depression, developmental speech/language disorders, intellectual disability, attention-deficit/hyperactivity disorder (ADHD), selective mutism, reactive attachment disorder, or childhood schizophrenia.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-12 (Estimated)

PRIMARY OUTCOMES:
Change in Total Score on the Childhood Autism Rating Scale (CARS) | Pre-FMT, 3 months post-FMT, and 6 months post-FMT
  The change from baseline to Week 24 in the total score of the Childhood Autism Rating Scale (CARS). The CARS is a 15-item behavioral rating scale used to diagnose and assess the severity of autism. Each item is scored from 1 to 4. The total score ranges from 15 to 60. A higher score indicates more severe autism symptoms.

SECONDARY OUTCOMES:
Change in Total Score on the Social Responsiveness Scale, Second Edition (SRS-2) | Pre-FMT, at Week 12, 24, and 48 post-FMT.
  Change from baseline to Weeks 12, 24, and 48. The SRS-2 assesses social impairments associated with autism spectrum disorders. Raw scores are converted to T-scores. Higher T-scores indicate greater severity of social impairment.
Change in Total Score on the Aberrant Behavior Checklist (ABC) | Pre-FMT, at Week 12, 24, and 48 post-FMT.
  Change from baseline to Weeks 12, 24, and 48. The ABC assesses problem behaviors in individuals with developmental disabilities. Higher scores indicate more severe problem behaviors.
Change in Total Score on the Gastrointestinal Symptom Rating Scale (GSRS) | Pre-FMT, during FMT, and at 2, 6, 12, 24, and 48 post-FMT.
  Change from baseline to Weeks 2, 6, 12, 24, and 48. The GSRS evaluates common gastrointestinal symptoms. Each item is scored from 1 (no discomfort) to 7 (very severe discomfort). Higher scores indicate worse GI symptoms.
Daily Stool Record (DSR) | Pre-FMT, during FMT, and at 2, 6, 12, 24 and 48 weeks post-FMT.
  Daily documentation of stool characteristics using the Bristol Stool Scale. The percentage of days with abnormal bowel movements (e.g., abnormal consistency, absence of stool, or use of GI medications) is calculated, with higher percentages indicating worse symptoms.
Change in Total Score on the Short Sensory Profile (SSP) | Pre-FMT, at12, 24 and 48 post-FMT.
  Change from baseline to Weeks 12, 24, and 48. The SSP measures sensory processing patterns in children. Lower scores indicate greater sensory processing difficulties.
Change in Total Score on the Children's Sleep Habits Questionnaire (CSHQ) | Pre-FMT, at12, 24 and 48 post-FMT.
  Change from baseline to Weeks 12, 24, and 48. The CSHQ assesses sleep problems in children. Higher scores indicate more disturbed sleep.
Change in Gut Microbiota Alpha Diversity (Shannon Index) | Pre-FMT, and at 2, 6, 12, 24 and 48 weeks post-FMT.
  Change from baseline to Weeks 2, 6, 12, 24, and 48 as measured by shotgun metagenomic sequencing. Alpha diversity measures the richness and evenness of microbial species within a sample.
Change in Relative Abundance of Specific Gut Microbial Taxa (at the genus level) | Pre-FMT, and at 2, 6, 12, 24 and 48 weeks post-FMT.
  Change from baseline to Weeks 2, 6, 12, 24, and 48 as measured by shotgun metagenomic sequencing (e.g., using MetaPhlAn for taxonomic profiling).
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From date of randomization until the end of study visit (Week 48).
  The number and percentage of participants experiencing any adverse event during the study period, graded for severity according to the Common Terminology Criteria for Adverse Events (CTCAE) v4.0. The relationship to the study intervention (FMT/placebo procedures) will be assessed by the investigator.
Incidence of Serious Adverse Events (SAEs) | From date of randomization until the end of study visit (Week 48).
  The number and percentage of participants experiencing any serious adverse event during the study period, as defined by CTCAE v4.0 and ICH guidelines.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Date for public release of raw data: within no later than 3 years after the publication of research results.
Access Criteria: To download data, contact must be made with the researcher.
URL: http://www.medresman.org.cn

REFERENCES:
- [Result] Ghirardini A, Nanni-Costa A, Venturi S, Ridolfi L, Petrini F, Taddei S, Venturoli A, Pugliese MR, Monti M, Martinelli G. Efficiency of organ procurement and transplantation programs. Transpl Int. 2000;13 Suppl 1:S267-71. doi: 10.1007/s001470050339. PMID 11112010
- [Result] Li Y, Xiao P, Ding H, Wang H, Xu Q, Wang R, Zheng L, Song X, Wang Y, Zhang T. Fecal Microbiota Transplantation in Children with Autism. Neuropsychiatr Dis Treat. 2024 Dec 9;20:2391-2400. doi: 10.2147/NDT.S488001. eCollection 2024. PMID 39677507
- [Result] Kang DW, Adams JB, Gregory AC, Borody T, Chittick L, Fasano A, Khoruts A, Geis E, Maldonado J, McDonough-Means S, Pollard EL, Roux S, Sadowsky MJ, Lipson KS, Sullivan MB, Caporaso JG, Krajmalnik-Brown R. Microbiota Transfer Therapy alters gut ecosystem and improves gastrointestinal and autism symptoms: an open-label study. Microbiome. 2017 Jan 23;5(1):10. doi: 10.1186/s40168-016-0225-7. PMID 28122648
- [Result] Chen K, Fu Y, Wang Y, Liao L, Xu H, Zhang A, Zhang J, Fan L, Ren J, Fang B. Therapeutic Effects of the In Vitro Cultured Human Gut Microbiota as Transplants on Altering Gut Microbiota and Improving Symptoms Associated with Autism Spectrum Disorder. Microb Ecol. 2020 Aug;80(2):475-486. doi: 10.1007/s00248-020-01494-w. Epub 2020 Feb 26. PMID 32100127
- [Result] Flora SJ, Tripathi N. Hepatic and renal metallothionein induction following single oral administration of gallium arsenide in rats. Biochem Mol Biol Int. 1998 Sep;45(6):1121-7. doi: 10.1080/15216549800203342. PMID 9762410
- [Result] Tan Q, Orsso CE, Deehan EC, Kung JY, Tun HM, Wine E, Madsen KL, Zwaigenbaum L, Haqq AM. Probiotics, prebiotics, synbiotics, and fecal microbiota transplantation in the treatment of behavioral symptoms of autism spectrum disorder: A systematic review. Autism Res. 2021 Sep;14(9):1820-1836. doi: 10.1002/aur.2560. Epub 2021 Jun 26. PMID 34173726
- [Result] Goncalves CL, Doifode T, Rezende VL, Costa MA, Rhoads JM, Soutullo CA. The many faces of microbiota-gut-brain axis in autism spectrum disorder. Life Sci. 2024 Jan 15;337:122357. doi: 10.1016/j.lfs.2023.122357. Epub 2023 Dec 19. PMID 38123016
- [Result] Ullah H, Arbab S, Tian Y, Chen Y, Liu CQ, Li Q, Li K. Crosstalk between gut microbiota and host immune system and its response to traumatic injury. Front Immunol. 2024 Jul 31;15:1413485. doi: 10.3389/fimmu.2024.1413485. eCollection 2024. PMID 39144142
- [Result] Njeh CF, Fuerst T, Diessel E, Genant HK, Hausler KD. Association between QUS and structural parameters? Calcif Tissue Int. 2000 Sep;67(3):273-4. doi: 10.1007/s002230001136. No abstract available. PMID 10954784
- [Result] Ullah H, Arbab S, Tian Y, Liu CQ, Chen Y, Qijie L, Khan MIU, Hassan IU, Li K. The gut microbiota-brain axis in neurological disorder. Front Neurosci. 2023 Aug 4;17:1225875. doi: 10.3389/fnins.2023.1225875. eCollection 2023. PMID 37600019
- [Result] Morton JT, Jin DM, Mills RH, Shao Y, Rahman G, McDonald D, Zhu Q, Balaban M, Jiang Y, Cantrell K, Gonzalez A, Carmel J, Frankiensztajn LM, Martin-Brevet S, Berding K, Needham BD, Zurita MF, David M, Averina OV, Kovtun AS, Noto A, Mussap M, Wang M, Frank DN, Li E, Zhou W, Fanos V, Danilenko VN, Wall DP, Cardenas P, Baldeon ME, Jacquemont S, Koren O, Elliott E, Xavier RJ, Mazmanian SK, Knight R, Gilbert JA, Donovan SM, Lawley TD, Carpenter B, Bonneau R, Taroncher-Oldenburg G. Multi-level analysis of the gut-brain axis shows autism spectrum disorder-associated molecular and microbial profiles. Nat Neurosci. 2023 Jul;26(7):1208-1217. doi: 10.1038/s41593-023-01361-0. Epub 2023 Jun 26. PMID 37365313
- [Result] You M, Chen N, Yang Y, Cheng L, He H, Cai Y, Liu Y, Liu H, Hong G. The gut microbiota-brain axis in neurological disorders. MedComm (2020). 2024 Jul 20;5(8):e656. doi: 10.1002/mco2.656. eCollection 2024 Aug. PMID 39036341
- [Result] O'Brien CP, Testa T, O'Brien TJ, Greenstein R. Conditioning in human opiate addicts. Pavlov J Biol Sci. 1976 Oct-Dec;11(4):195-202. doi: 10.1007/BF03000314. PMID 995439
- [Result] Kodak T, Bergmann S. Autism Spectrum Disorder: Characteristics, Associated Behaviors, and Early Intervention. Pediatr Clin North Am. 2020 Jun;67(3):525-535. doi: 10.1016/j.pcl.2020.02.007. Epub 2020 May 4. PMID 32443991
- [Result] Penel C, Greppin H. Binding of plant isoperoxidases to pectin in the presence of calcium. FEBS Lett. 1994 Apr 18;343(1):51-5. doi: 10.1016/0014-5793(94)80605-5. PMID 8163016
- [Result] Sundkvist T. Impact of postmenopausal hormone therapy on cardiovascular events and cancer. Combining thromboembolic events with cardiovascular events does not support odds ratio of 0.7. BMJ. 1997 Sep 13;315(7109):677. No abstract available. PMID 9310578
- [Result] Senti M, Puig JM, Lloveras J, Aubo C, Mir M, Barbosa F, Oliveras A, Masramon J. Effect of cyclosporine on serum lipoprotein(a) levels in renal transplant recipients. Transplant Proc. 1997 Aug;29(5):2404-5. doi: 10.1016/s0041-1345(97)00421-1. No abstract available. PMID 9270782
- [Result] Bentele MJ, Vig KW, Shanker S, Beck FM. Efficacy of training dental students in the index of orthodontic treatment need. Am J Orthod Dentofacial Orthop. 2002 Nov;122(5):456-62. doi: 10.1067/mod.2002.126895. PMID 12439472
- [Result] Hirota T, King BH. Autism Spectrum Disorder: A Review. JAMA. 2023 Jan 10;329(2):157-168. doi: 10.1001/jama.2022.23661. PMID 36625807

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT07381374/Prot_SAP_002.pdf
  • Informed Consent Form (2025-03-19): https://cdn.clinicaltrials.gov/large-docs/74/NCT07381374/ICF_001.pdf